CLINICAL TRIAL: NCT03988348
Title: Perioperative Outcome of Infraumbilical Versus a Modified Intraumbilical Direct Trocar Insertion in Gynecologic Laparoscopy: A Randomized Controlled Trial
Brief Title: Perioperative Outcome of Infraumbilical Versus a Modified Intraumbilical Direct Trocar Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUL
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): infraumbilical transverse incision will be done
  Interventions: Procedure: infraumbilical transverse incision
- control group (Active Comparator): Direct intraumbilical transverse incision will be done
  Interventions: Procedure: intraumbilical incision

INTERVENTIONS:
Procedure: infraumbilical transverse incision — a 10 mm infraumbilical transverse incision will be done to allow trocar to be inserted without undue resistance from the skin so that the trocar will pass through the fascia and the peritoneum with ease
  Arms: study group
Procedure: intraumbilical incision — right sided curved longitudinal intraumbilical incision will be performed for initial intraperitoneal access
  Arms: control group

SUMMARY:
Laparoscopic surgery is now a well-established alternative to open surgery for many gynecological disorders owing to its faster wound healing, shorter hospital stay, less postoperative pain, and better cosmetic results. Postoperative scar cosmoses is a critical issue for women, especially for young women. These scars may have negative impacts, such as psychological consequences. The symptoms associated with the wound, such as pain, tenderness, and itching, can be induced by the scars

ELIGIBILITY:
Inclusion Criteria:

* All women subjected to direct trocar application as a part of any gynecologic procedure performed

Exclusion Criteria:

* Verres needle insertion.
* Patients with previous abdominal surgery and scar,
* umbilical hernia,
* previous laparoscopy or previous umbilical surgery,
* burns in the umbilical region;
* who have hyperpigmented skins.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-08-04 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
the mean difference in the duration of surgery | 30 minutes
  calculated from the onset of surgery till the end

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt